CLINICAL TRIAL: NCT04308239
Title: Reactive Balance Training Targeting Both Slip- and Trip-Induced Falls Among Older Adults: a Pilot Randomized Controlled Trial
Brief Title: Reactive Balance Training Targeting Both Slip- and Trip-Induced Falls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Michael Madigan, Professor, Virginia Polytechnic Institute and State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-486
Record Dates: First submitted 2020-03-04; First posted 2020-03-16 (Actual); Results first posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-03

CONDITIONS: Accidental Fall
Keywords: balance training; step training; perturbation-based balance training; dynamic balance; aging

STUDY DESIGN:
Intervention Model Description: A two-group, pretest-posttest parallel design was employed. Participants were first assigned to either the reactive balance training or control intervention using minimization. During the first week, participants completed a pre-intervention assessment involving exposure to a single laboratory-induced slip or trip based upon random assignment. During the second and third weeks, participants completed a total of four sessions of their assigned intervention (two sessions per week for two weeks). During the fourth week, participants completed a post-intervention assessment involving exposure to the other perturbation (slip or trip) that they did not experience during the pre-intervention assessment. This design was selected to evaluate gait and reactive balance prior to any training intervention, and to avoid any unintended training effects induced by exposing participants to the same perturbation more than once.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reactive balance training (Experimental): Four training sessions, conducted twice a week for two weeks in groups of 1-2 participants. Each session was 0.5-1 hours, with an active training time of 30 minutes for each participant.
  Reactive balance training involved both slip and trip training.
  Slip training involved repeatedly stepping onto a low-friction interface (nylon fabric placed over a 0.9 × 0.9 meter polycarbonate sheet) while practicing controlling/decelerating the slipping foot and properly positioning the non-slipping foot under the pelvis.
  Trip training involved repeatedly practicing recovery from simulated trips on a modified treadmill. While standing on a modified treadmill, the treadmill belt was quickly accelerated posteriorly to elicit a forward loss of balance that mimicked a trip while walking. Participants attempted to step to avert a fall, and to establish a stable gait on the treadmill, after which the treadmill speed was slowed to zero to complete the trial.
  Interventions: Behavioral: Reactive balance training
- Control balance training (Active Comparator): Four training sessions, conducted twice a week for two weeks in groups of 1-2 participants. Each session was 0.5-1 hours, with an active training time of 30 minutes for each participant.
  The control intervention involved general balance exercises adapted from the Otago Exercise program. Briefly, all four sessions involved balance exercises and strength exercises using ankle weights, and were progressively increased as performance improved by increasing ankle weights or the difficulty of the balance exercises (e.g., not holding onto a wall or support).
  Interventions: Behavioral: Otago Balance Training

INTERVENTIONS:
Behavioral: Reactive balance training — Participants were exposed to simulated trips and slips under safe, controlled conditions in order to practice their reactive response to these common balance perturbations.
  Arms: Reactive balance training
Behavioral: Otago Balance Training — Balance exercises and strength exercises using ankle weights, and were progressively increased as performance improved by increasing ankle weights or the difficulty of the balance exercises (e.g., not holding onto a wall or support).
  Arms: Control balance training

SUMMARY:
The goal of this study was to evaluate the effects of reactive balance training (RBT) targeting slipping and tripping on laboratory-induced slips and trips. In an effort to build upon prior work, the present study included: 1) a control group receiving an alternative balance training intervention; 2) separate training and assessment sessions; 3) alternative RBT methods that may be more amenable to work outside the lab compared to prior methods, and 4) older adult participants receiving individualized training to reduce drop-out. The investigators hypothesized that slips after RBT would result in improved reactive balance kinematics, and a lower incidence of falls, compared to either initial slips before any intervention or after a control intervention. The investigators also hypothesized that trips after RBT would result in improved reactive balance kinematics, and a lower incidence of falls, compared to either initial trips before any intervention or after a control intervention. Results were intended to contribute to knowledge regarding the efficacy of alternative methods for RBT, and provide additional evidence regarding its efficacy.

ELIGIBILITY:
Inclusion Criteria:

1) pass a medical history and screening administered by a physician that excluded participants with osteoporosis of the lumbar spine or proximal femur as assessed by Dual Energy X-ray Absorptiometry (Lunar iDXA, GE Healthcare, Chicago, IL), or any unstable or progressive medical conditions that could contribute to imbalance or falls

Exclusion Criteria:

1. smoked
2. were in physical therapy
3. had a self-reported fragility fracture within the last 10 years
4. had an acute lower extremity injury within the last 3 months
5. had lower extremity surgery within the last six months
6. had an ankle arthroplasty
7. had a knee or hip arthroplasty within the last 12 months

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Madigan, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech - Department of Industrial and Systems Engineering, Blacksburg, Virginia, United States

REFERENCES:
- [Derived] Allin LJ, Brolinson PG, Beach BM, Kim S, Nussbaum MA, Roberto KA, Madigan ML. Perturbation-based balance training targeting both slip- and trip-induced falls among older adults: a randomized controlled trial. BMC Geriatr. 2020 Jun 12;20(1):205. doi: 10.1186/s12877-020-01605-9. PMID 32532221

RESULTS

PARTICIPANT FLOW:
Groups:
- Reactive Balance Training: Four training sessions, conducted twice a week for two weeks in groups of 1-2 participants. Training in each session was 30 minutes for each participant.
  Reactive balance training involved both slip and trip training.
  Slip training involved repeatedly stepping onto a low-friction interface (nylon fabric placed over a 0.9 × 0.9 meter polycarbonate sheet) while practicing controlling/decelerating the slipping foot and properly positioning the non-slipping foot under the pelvis.
  Trip training involved repeatedly practicing recovery from simulated trips on a modified treadmill. While standing on a modified treadmill, the treadmill belt was quickly accelerated posteriorly to elicit a forward loss of balance that mimicked a trip while walking. Participants attempted to step to avert a fall, and to establish a stable gait on the treadmill, after which the treadmill speed was slowed to zero to complete the trial.
- Control Balance Training: Four training sessions, conducted twice a week for two weeks in groups of 1-2 participants. Each session was 0.5-1 hours, with an active training time of 30 minutes for each participant.
  The control intervention involved general balance exercises adapted from the Otago Exercise program. Briefly, all four sessions involved balance exercises and strength exercises using ankle weights, and were progressively increased as performance improved by increasing ankle weights or the difficulty of the balance exercises (e.g., not holding onto a wall or support).
  Otago Balance Training: Balance exercises and strength exercises using ankle weights, and were progressively increased as performance improved by increasing ankle weights or the difficulty of the balance exercises (e.g., not holding onto a wall or support).
Period: Pre-intervention Evaluation (1 Week)
Arm/Group | Reactive Balance Training | Control Balance Training
Started | 20 | 14
Completed | 17 (No withdrawals. These participants just missed this evaluation but stayed in study.) | 11 (No withdrawals. These participants just missed this evaluation but stayed in study.)
Not Completed | 3 | 3
Not completed — Did not attend due to schedule conflict | 2 | 1
Not completed — testing error during evaluation | 1 | 2
Period: Intervention (2 Weeks)
Arm/Group | Reactive Balance Training | Control Balance Training
Started | 20 | 14
Completed | 20 | 14
Not Completed | 0 | 0
Period: Post-intervention Evaluation (1 Week)
Arm/Group | Reactive Balance Training | Control Balance Training
Started | 20 | 14
Completed | 19 | 10
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — testing error during evaluation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Reactive Balance Training: Group of participants who were assigned to reactive balance training.
- Control Balance Training: Group of participants who were assigned to control balance training.
- Total: Total of all reporting groups
Arm/Group | Reactive Balance Training | Control Balance Training | Total
Number analyzed (Participants) | 20 | 14 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (4.4) | 70.0 (4.0) | 69.3 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 9 | 6 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Mass [Mean (Standard Deviation); unit: kilograms] | 77.8 (15.5) | 80.0 (14.7) | 78.7 (15.0)

OUTCOME MEASURES:

1. Primary Outcome: Peak Slip Speed
Description: highest instantaneous speed of slipping foot during actual slip
Time Frame: during week 1, before the intervention that spanned weeks 2 and 3
Measure: Mean (Standard Deviation); unit: meters/sec
Groups:
- Baseline SLIP Group: Group of participants who were slipped prior to intervention.
Arm/Group | Baseline SLIP Group
Number analyzed (Participants) | 11
meters/sec | 2.8 (.32)

2. Primary Outcome: Peak Slip Speed
Description: highest instantaneous speed of slipping foot during actual slip
Time Frame: during week 4, after the intervention that spanned weeks 2 and 3
Measure: Mean (Standard Deviation); unit: meters/sec
Groups:
- Post-Control Balance Training SLIP Group: Group of participants who were slipped after the control balance training intervention.
- Post-Reactive Balance Training SLIP Group: Group of participants who were slipped after the reactive balance training intervention.
Arm/Group | Post-Control Balance Training SLIP Group | Post-Reactive Balance Training SLIP Group
Number analyzed (Participants) | 5 | 11
meters/sec | 3.15 (.33) | 2.58 (.41)

3. Primary Outcome: Trunk Angle at Touchdown After Tripping
Description: anterior-posterior trunk angle relative to vertical at instant of touchdown of initial recovery step over tripping obstacle
Time Frame: during week 1, before the intervention that spanned weeks 2 and 3
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Baseline TRIP Group: Group of participants who were tripped prior to intervention.
Arm/Group | Baseline TRIP Group
Number analyzed (Participants) | 17
degrees | 37 (9.6)

4. Primary Outcome: Trunk Angle at Touchdown After Tripping
Description: as for outcome 3
Time Frame: during week 4, after the intervention that spanned weeks 2 and 3
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Post-Control Balance Training TRIP Group: Group of participants who were tripped after the control balance training intervention.
- Post-Reactive Balance Training TRIP Group: Group of participants who were tripped after the reactive balance training intervention.
Arm/Group | Post-Control Balance Training TRIP Group | Post-Reactive Balance Training TRIP Group
Number analyzed (Participants) | 5 | 8
degrees | 36.9 (2.2) | 41.1 (3.7)

5. Secondary Outcome: Slip Distance
Description: distance moved by slipping foot during actual slip
Time Frame: during week 1, before the intervention that spanned weeks 2 and 3
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Baseline SLIP Group
Number analyzed (Participants) | 11
centimeters | 80.8 (4.5)

6. Secondary Outcome: Slip Distance
Description: distance moved by slipping foot during actual slip
Time Frame: during week 4, after the intervention that spanned weeks 2 and 3
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Post-Control Balance Training SLIP Group | Post-Reactive Balance Training SLIP Group
Number analyzed (Participants) | 5 | 11
centimeters | 74.2 (6.6) | 71.4 (4.5)

7. Secondary Outcome: Fall Incidence After a Laboratory-induced Slip
Description: the outcome of each slip was categorized as either a: fall, recovery, or harness-assisted
Time Frame: during week 1, before the intervention that spanned weeks 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline SLIP Group
Number analyzed (Participants) | 10
Participants | 8

8. Secondary Outcome: Fall Incidence After a Laboratory-induced Slip
Description: the outcome of each slip was categorized as either a: fall, recovery, or harness-assisted
Time Frame: during week 4, after the intervention that spanned weeks 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Control Balance Training SLIP Group | Post-Reactive Balance Training SLIP Group
Number analyzed (Participants) | 5 | 11
Participants | 3 | 2

9. Secondary Outcome: Recovery Step Length After Tripping
Description: anterior-posterior step distance of first step over tripping obstacle
Time Frame: during week 1, before the intervention that spanned weeks 2 and 3
Measure: Mean (Standard Deviation); unit: percent body height
Arm/Group | Baseline TRIP Group
Number analyzed (Participants) | 17
percent body height | 54.3 (14.1)

10. Secondary Outcome: Recovery Step Length After Tripping
Description: anterior-posterior step distance of first step over tripping obstacle
Time Frame: during week 4, after the intervention that spanned weeks 2 and 3
Measure: Mean (Standard Deviation); unit: percent body height
Arm/Group | Post-Control Balance Training TRIP Group | Post-Reactive Balance Training TRIP Group
Number analyzed (Participants) | 5 | 8
percent body height | 53.7 (8.8) | 64.1 (10.5)

11. Secondary Outcome: Fall Incidence After a Laboratory-induced Trip
Description: the outcome of each trip was categorized as a: fall, recovery, or harness-assisted
Time Frame: during week 1, before the intervention that spanned weeks 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline TRIP Group
Number analyzed (Participants) | 17
Participants | 6

12. Secondary Outcome: Fall Incidence After a Laboratory-induced Trip
Description: the outcome of each trip was categorized as a: fall, recovery, or harness-assisted
Time Frame: during week 4, after the intervention that spanned weeks 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Control Balance Training TRIP Group | Post-Reactive Balance Training TRIP Group
Number analyzed (Participants) | 5 | 8
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: The period of time over which adverse event data were collected was 4 weeks. This included week 1 of pre-intervention evaluation, weeks 2-3 of intervention, and week 4 of post-intervention evaluation.
Groups:
- Reactive Balance Training: Participants assigned to the reactive balance training.
- Control Balance Training: Participants assigned to the control balance training.
Arm/Group | Reactive Balance Training | Control Balance Training
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/5
Other Adverse Events (participants affected / at risk) | 1/11 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reactive Balance Training (N=11) | Control Balance Training (N=5)
Baker's cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not believed to have resulted from reactive balance training or testing involved in this study.
Arthritis pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
All training and assessment sessions were conducted by a single investigator who was not blinded to participant group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT04308239/Prot_SAP_ICF_000.pdf